CLINICAL TRIAL: NCT07314775
Title: Yangxin Dawayimixike Honey Paste for Carotid Atherosclerotic Plaque With Dyslipidemia: A Randomized Controlled Clinical Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xinjiang Uygur Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024ZD0528302
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dyslipidemia; Carotid Atherosclerotic Plaques
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Yangxin Dawayimixike Honey Paste placebo
- Yangxin Dawayimixike Honey Paste (Experimental)
  Interventions: Drug: Yangxin Dawayimixike Honey Paste

INTERVENTIONS:
Drug: Yangxin Dawayimixike Honey Paste — 3 g bid po
  Arms: Yangxin Dawayimixike Honey Paste
Drug: Yangxin Dawayimixike Honey Paste placebo — 3 g bid po
  Arms: Placebo

SUMMARY:
This clinical trial aims to evaluate the efficacy and safety of Yangxin Dawayimixike Honey Paste in intervening carotid atherosclerotic plaque combined with dyslipidemia. The study will enroll patients with carotid atherosclerotic plaque and dyslipidemia in a multicenter, randomized, double-blind, placebo-controlled trial. Based on standardized Western medical treatment, the treatment group will receive Yangxin Dawayimixike Honey Paste, while the control group will receive a simulated preparation of Yangxin Dawayimixike Honey Paste. The treatment duration is 12 months, followed by a one-year follow-up period.

The primary efficacy endpoint is the change in intima-media thickness (IMT) of the carotid artery. Secondary efficacy endpoints include plaque Crouse score, plaque area, vascular remodeling index (RI), major adverse cardiovascular events (MACE), four lipid parameters (total cholesterol, triglycerides, LDL-C, HDL-C), Traditional Chinese Medicine syndrome score, and quality of life scale (SF-36). Safety indicators include vital signs (respiration, pulse, heart rate, blood pressure), complete blood count, routine urinalysis, routine stool examination, liver and kidney function tests, and four coagulation parameters. These measures will be used to assess the treatment's efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for Carotid Atherosclerotic Plaque (CAP);
2. Meets the diagnostic criteria for dyslipidemia;
3. Meets the TCM syndrome differentiation criteria for Qi Stagnation and Blood Stasis pattern;
4. Aged 18-75 years, both sexes eligible;
5. Vital signs stable, conscious with normal communication ability;
6. Subject voluntarily participates and signs the informed consent form.

Exclusion Criteria:

1. Patients with severe cardiovascular diseases, including acute myocardial infarction, unstable angina, NYHA Class II-IV heart failure, severe arrhythmias, congenital heart disease, or severe valvular heart disease;
2. Patients with poorly controlled hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure >100 mmHg), severe cerebrovascular diseases, hemorrhagic or hematologic disorders, or malignant tumors;
3. Patients with hepatic dysfunction, defined as alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels exceeding twice the upper limit of normal, or renal insufficiency, defined as serum creatinine levels exceeding 1.5 times the upper limit of normal;
4. Patients with severe psychological disorders, intellectual disabilities, or language barriers;
5. Pregnant or lactating women;
6. Patients with known hypersensitivity to the investigational drug;
7. Patients concurrently participating in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
carotid intima-media thickness | 12 months

SECONDARY OUTCOMES:
Plaque Crouse Score | 12 months
plaque area | 12 months
RI (Vascular Remodeling Index) | 12 months
MACE (Major Adverse Cardiovascular Events) | 12 months
total cholesterol, triglycerides, LDL-C, HDL-C | 12 months
Traditional Chinese Medicine syndrome score | 12 months
36-Item Short Form Health Survey | 12 months
24-item Hamilton Depression Rating Scale | 12 months
14-item Hamilton Anxiety Rating Scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sun Longfei Sun Longfei, Ph.D., Principal Investigator — Xinjiang Uygur Autonomous Region Traditional Chinese Medicine Hospital

IPD SHARING:
Plan to Share IPD: Undecided